CLINICAL TRIAL: NCT06075524
Title: Maximizing Anti-PD-1 Therapy by Monitoring T Cell Responses in Melanoma, Lung and Other Cancer Types
Brief Title: Evaluation of Anti-PD-1 Therapy by Monitoring T Cell Responses in Melanoma, Lung and Other Cancer Types
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC200706; NCI-2022-08127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-000934 (Other: Mayo Clinic Institutional Review Board); MC200706 (Other: Mayo Clinic in Rochester); F30CA250326 (NIH); R21CA197878 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Locally Advanced Lung Carcinoma; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Melanoma; Metastatic Lung Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Melanoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from the blood and stool specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Blood and stool sample collection): Patients undergo blood sample collection throughout the study. Patients also undergo optional stool sample collection and have their medical records reviewed on study. In addition, patients provide previously-collected tissue sample, if available.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and optional stool/tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study explores the role of T cells in monitoring disease status and response during anti-PD-1/PD-L1 treatment in patients with melanoma, lung and other cancer types. Measuring levels of specific targets such as Bim and soluble PD-L1 during therapy may help track treatment resistance and clinical outcomes. This information may also help researchers determine why some people with melanoma, lung and other cancer types respond to PD-1/PD-L1 treatment and others do not.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the role of Bim for monitoring disease status during anti-PD-1 therapy.

II. Identify the mechanisms of resistance to anti-PD-1 blockade. III. Quantify and modulate levels of NKG7 messenger ribonucleic acid (mRNA) in CD8+ T cells.

OUTLINE: This is an observational study.

Patients undergo blood sample collection throughout the study. Patients also undergo optional stool sample collection and have their medical records reviewed on study. In addition, patients provide previously-collected tissue sample, if available.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Have histologic evidence of locally or regionally advanced or stage IV malignancy
* Are considered appropriate for starting therapy with anti-PD-1/anti-PD-L1 monoclonal antibody by their treating physician (prior therapy with immune checkpoint inhibitor (ICI) is allowed)
* Have an understanding of the protocol and its requirements, risks, and discomforts
* Are willing to undergo peripheral blood collection at the time points mentioned in the protocol
* Are able and willing to sign an informed consent

Exclusion Criteria:

* Inability on the part of the patient to understand the informed consent or be compliant with the protocol
* Patients receiving any concurrent anti-cancer therapy or investigational agents (with the exception of an anti-PD-1/anti-PD-L1 agent as mentioned above)
* Patients who are pregnant, nursing, or are of childbearing potential and are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma, lung or other cancer recruited from the clinical practice in the Department of Oncology at Mayo Clinic in Rochester, Minnesota who are considered appropriate for starting therapy with an open-label commercially available, FDA approved anti-PD-1 monoclonal antibody by their treating provider.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Role of Bim for monitoring disease status during anti-PD-1 therapy | Up to 10 samples: at baseline; 6 weeks after initiation of therapy; subsequently at each radiographic tumor assessment (starting at approx. 9-12 weeks) including at confirmed disease progression.
  Will be assessed by serial measurements of Bim levels in tumor-reactive CD8+ T cells from the peripheral blood of patients with advanced cancer undergoing therapy with an anti-PD-1 monoclonal antibody and correlate them with clinical outcome.
Mechanisms of resistance to anti-PD-1 blockade | Up to 10 samples: at baseline; 6 weeks after initiation of therapy; subsequently at each radiographic tumor assessment (starting at approx. 9-12 weeks) including at confirmed disease progression.
  Will be assessed by reviewing blood samples to determine whether high sPD-L1 levels are associated with higher Bim levels in CD11ahigh PD-1+CD8+ T cells and decreased response to single-agent anti-PD1 blocking antibody in patients with cancer.
Quantify and modulate levels of NKG7 mRNA in CD8+ T cells | Up to 10 samples: at baseline; 6 weeks after initiation of therapy; subsequently at each radiographic tumor assessment (starting at approx. 9-12 weeks) including at confirmed disease progression.
  CD8+ T cells will be isolated from the peripheral blood of patients with advanced cancer, and messenger ribonucleic acid (mRNA) will be isolated. Qualitative and quantitative reverse transcription polymerase chain reaction (RT-PCR) assays will be performed on these samples in order to determine the levels of six different mRNA splice variants of NKG7. Results will be compared to clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir N. Markovic, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials